CLINICAL TRIAL: NCT04281407
Title: Impact of Probiotics on Drug, Vitamin, and Hormone Metabolism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Yvonne Lin, Associate Professor: Department of Pharmaceutics, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00007095
Record Dates: First submitted 2020-02-11; First posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Metabolism
Keywords: drug metabolism; CYP3A; UGT; SULT

STUDY DESIGN:
Intervention Model Description: Single arm prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probiotics treatment on midazolam and acetaminophen metabolism (Experimental): Experimental:
  Day 1: midazolam (2 mg oral) + acetaminophen (500 mg oral) + midazolam (1 mg IV) Days 1-28: Visbiome (2 capsules) administered BID Day 11: midazolam (2 mg oral) + acetaminophen (500 mg oral) + midazolam (1 mg IV)
  Interventions: Dietary Supplement: Visbiome

INTERVENTIONS:
Dietary Supplement: Visbiome — 2 capsules of Visbiome, a probiotics supplement, twice a day (morning and evening) for 28 days

SUMMARY:
This is an open-label, fixed sequence study of the effect of probiotics supplementation on drug, vitamin, and hormone metabolism.

DETAILED DESCRIPTION:
The investigators hypothesize that probiotic treatment (Visbiome) will alter the activities of major classes of drug metabolizing enzymes. Twelve healthy male subjects will participate in a pharmacokinetic study prior to and following supplementation with Visbiome probiotics for 28 days.

The investigators will determine the pharmacokinetics of oral and intravenous midazolam [metabolized by cytochrome P450 3A enzymes, uridine 5'-diphospho-glucuronosyltransferases (UGTs) and sulfotransferase (SULTs)] and acetaminophen (metabolized by UGTs and SULTs), and the circulating concentrations of endogenous compounds (i.e., testosterone and vitamin D metabolites) prior to and following supplementation with Visbiome probiotics for 28 days. In addition, the investigators will compare the fecal microbiota composition and plasma lipidomic and metabolomics profiles to assess the impact of Visbiome supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 to 40 years old.
* Biological male participants only with no preference to ethnicity. Women are excluded as one of the aims is to determine the impact of probiotics supplementation on testosterone metabolism. As testosterone and metabolite levels are higher in men than in women, men will be recruited to have an increased ability to detect a difference.
* Have a body mass index between 25 and 3218.5 and 27 kg/m2.
* Be currently in good health without a self-reported history of liver, kidney, gastrointestinal or heart disease, and within the normal range or up to 15% of the upper end of the reference range on the Comprehensive and Hepatic Panel.
* Participants must agree to take 2 capsules of Visbiome, a probiotics supplement provided by the study coordinators, twice a day (morning and evening) from Study Day 2 to 29.
* Participants must agree not to take any prescription drugs for the entire duration of the study. This list includes, but is not restricted to, azole antifungal agents, macrolide antibiotics, anti-seizure medications, antihypertensive agents, cholesterol lowering agents, retinoids, corticosteroids, or immunosuppressant medications for the duration of the study.
* Participants must be willing to avoid ingesting grapefruit, grapefruit juice or other grapefruit juice containing products during the study.
* If an over-the-counter medication is needed, the participant should contact the study coordinator for verification and upon approval, the OTCs can be taken but should not be used 24 hours before each study visit and during the study visits.
* Willing to fast overnight before the pharmacokinetic study days.
* Willing to abstain from alcohol-containing beverages 24 hours before and during the study visits.

Exclusion Criteria:

* Milk allergy or lactose intolerance.
* Currently using prescription medications. Participants may participate in the study following a 2-week washout after discontinuing any prescription medication upon approval of the study team.
* Current cigarette smoker.
* Individuals with systemic disorders affecting the immune system (e.g., HIV, connective tissue disorders, cancers, etc.)
* Self-reported history of liver, kidney, gastrointestinal (e.g., Ulcerative Colitis or Crohn's Disease, intestinal stricture, stenosis, obstruction, fistula, abscess, or ileostomy) or heart disease.
* Abnormal liver or kidney function tests based on the Comprehensive and Hepatic Panel (below the lower end or greater than 15% of the upper end of the reference range).
* Known or suspected history of alcohol or drug abuse.
* Allergic to midazolam, triazolam, diazepam, or lorazepam.
* Recent ingestion (<1 week) of any medication known to be metabolized by CYP3A4 or alter CYP3A activity.
* Unable to give informed consent.
* Participated in another clinical trial or study within 30 days.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-01-03 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Oral midazolam peak concentration (Cmax) | 0 to 3 hours on Days 1 and 29
  Following 2 mg midazolam syrup given orally at time = 0
IV midazolam peak concentration (Cmax) | 3 to 12 hours on Days 1 and 29
  Following 1 mg midazolam given IV at time = 3 hrs
Overall midazolam area under the curve (AUC) | 0 to 12 hours on Days 1 and 29
  Following 2 mg midazolam syrup given orally and 1 mg midazolam given IV
Overall 1'-hydroxymidazolam area under the curve (AUC) | 0 to 12 hours on Days 1 and 29
  Following 2 mg midazolam syrup given orally and 1 mg midazolam given IV
Acetaminophen peak concentration (Cmax) | 0 to 12 hours on Days 1 and 29
  500 mg acetaminophen given orally
Acetaminophen area under the curve (AUC) | 0 to 12 hours on Days 1 and 29
  500 mg acetaminophen given orally at time = 0
Acetaminophen-glucuronide area under the curve (AUC) | 0 to 12 hours on Days 1 and 29
  500 mg acetaminophen given orally at time = 0
Acetaminophen-sulfate area under the curve (AUC) | 0 to 12 hours on Days 1 and 29
  500 mg acetaminophen given orally at time = 0

SECONDARY OUTCOMES:
Midazolam terminal half-life | 0 to 12 hours on Days 1 and 29
  Following 2 mg midazolam syrup given orally and 1 mg midazolam given IV
Acetaminophen terminal half-life | 0 to 12 hours on Days 1 and 29
  500 mg acetaminophen given orally at time = 0
Urinary excretion of 1'-hydroxymidazolam | 0 to 12 hours on Days 1 and 29
  Amount of 1'-hydroxymidazolam recovered in urine
Urinary excretion of acetaminophen-glucuronide | 0 to 12 hours on Days 1 and 29
  Amount of acetaminophen-glucuronide recovered in urine
Urinary excretion of acetaminophen-sulfate | 0 to 12 hours on Days 1 and 29
  Amount of acetaminophen-sulfate recovered in urine

OTHER OUTCOMES:
Microbiome composition of fecal sample | Days 1 and 29
  Compositional studies using sequencing of 16S gene

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Lin, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States